CLINICAL TRIAL: NCT05380193
Title: Serotype Distribution in Hospitalized Adult With Pneumococcal Community Acquired Pneumonia in France
Acronym: CAP'Hospi
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C21-24; 2021-A03157-34 (Registry Identifier: ID RCB)
Record Dates: First submitted 2022-03-07; First posted 2022-05-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pneumonia; Pneumococcal Infections; Community-acquired Pneumonia
Keywords: France; Vaccine; pneumococcal infections
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CAP'Hospi is an observational, multicentric study in France which primary objective is to describe the proportion of Community Acquired Pneumonia due to serotypes included in PCV20 among adults hospitalized for CAP

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older
2. Admission to hospital for at least 24 hours
3. Suspicion of community-acquired pneumonia at admission defined as the association of: Radiologic findings consistent with pneumonia (eg, pleural effusion, increased pulmonary density due to infection and/or alveolar infiltrates [multilobar, lobar, or segmental] containing air bronchograms), AND The presence of ≥2 of the following signs or symptoms: Fever (oral temperature >38°C or tympanic temperature >38.5°C) in the 24 hours preceding admission; Hypothermia (<35.5°C measured by a healthcare provider) in the 24 hours preceding admission ; Chills or rigors ; Pleuritic chest pain ; New or worsening cough ; Sputum production ; Dyspnea (shortness of breath); Tachypnea (respiratory rate >20/min) ; Malaise ; Abnormal auscultatory findings suggestive of pneumonia (rales or evidence of pulmonary consolidation)
4. Written informed consent from the patient

Exclusion Criteria:

1. Suspicion of tuberculosis
2. Individuals placed under judicial protection
3. Individuals who refuse the transfer of biological samples to the USA
4. Patient developing signs and symptoms of pneumonia after having been hospitalized for 48 hours or more
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults hospitalized more than 24h for Community Acquired Pneumonia
Sampling Method: Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
proportions of S. pneumoniae serotypes included in PCV20 | 2 years
  The proportion will be determined by UAD assay and/or culture from any sites overall and by age and risk group among adults hospitalized with CAP

SECONDARY OUTCOMES:
proportion of serotypes of S. pneumoniae by group | 2 years
  Among adults hospitalized for all-cause CAP or pneumococcal CAP the proportion of serotypes of S. pneumoniae grouped by serotypes included into pneumococcal vaccines and individual serotypes, by age and risk group
Patients hospital trajectories | 2 years
  The proportion of patients who died from any cause, the proportion of patients requiring mechanical ventilation within the first 30 days of hospitalization, the proportion of patients who required transfer to ICU within the first 30 days of hospitalization, the length of ICU-stay, the length of hospital-stay, the proportion of patients who required hospital re-admission
Patients hospital stay by serotype groups | 2 years
  The proportion of patients who died from any cause, the proportion of patients requiring mechanical ventilation within the first 30 days of hospitalization, the proportion of patients who required transfer to ICU within the first 30 days of hospitalization, the length of ICU-stay, the length of hospital-stay, the proportion of patients who required hospital re-admission
Prevalence of different bacterial and viral causes of hospitalized CAP | 2 years
  description of the proportion of bacteria and virus attributable to each patients
The proportion of patients with a severe CAP | 2 years
  transfer to the ICU during hospitalization. Studied factors will include baseline characteristics of patients and pneumococcal and pneumococcal serotype pneumonia etiology
The proportion of patients who required re-hospitalization following hospital discharge | 2 years
  Studied factors will include baseline characteristics of patients and pneumococcal and pneumococcal serotype pneumonia etiology

CONTACTS AND LOCATIONS:
Overall Officials: Liem B Luong, MD, Principal Investigator — CIC 1417 Cochin-Pasteur
Locations (5):
- France (5):
  - CHU Rennes, Rennes, Brittany Region
  - Hopital de la Croix Rousse, Hospices Civils de Lyon, Lyon
  - Hôpital Cochin, Paris
  - Hôpital Bichat, Paris
  - CHU de Saint-Etienne, Saint-Etienne